CLINICAL TRIAL: NCT05175300
Title: Interest of a Highly Cross-linked Polyethylene Acetabular Component Doped With Vitamin E in Total Hip Arthroplasty of the Young and Active Subject
Acronym: ICARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-A02040-41
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hip Arthropathy
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: A single-centre, prospective, randomised, single-blind, comparative, category 2 study of two parallel groups of patients undergoing total hip arthroplasty:
  * Group 1: Prosthesis with a second-generation ceramic-on-highly cross-linked polyethylene (CoPXE) couple.
  * Group 2: Prosthesis with ceramic-on-ceramic (CoC) torque.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Prosthesis with a second-generation ceramic-on-highly cross-linked polyethylene (CoPXE) couple.
  Interventions: Device: Prosthesis with CoPXE couple.
- Group 2 (Active Comparator): Prosthesis with ceramic-on-ceramic (CoC) torque.
  Interventions: Device: Prosthesis with CoC torque.

INTERVENTIONS:
Device: Prosthesis with CoPXE couple. — Prosthesis with a second-generation ceramic-on-highly cross-linked polyethylene (CoPXE) couple.
  Arms: Group 1
Device: Prosthesis with CoC torque. — Prosthesis with ceramic-on-ceramic (CoC) torque.
  Arms: Group 2

SUMMARY:
Interest of a highly cross-linked polyethylene acetabular component doped with vitamin E in total hip arthroplasty of the young and active subject.

DETAILED DESCRIPTION:
A single-centre, prospective, randomised, single-blind, comparative study of two parallel groups of patients undergoing total hip arthroplasty:

* Group 1: Prosthesis with a second-generation ceramic-on-highly cross-linked polyethylene (CoPXE) couple.
* Group 2: Prosthesis with ceramic-on-ceramic (CoC) torque.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 65 years,
* Who have signed their consent to participate in the study,
* For whom an indication for total hip arthroplasty has been given

Exclusion Criteria:

* History of hip surgery
* Indication for a dual mobility prosthesis (obese patient, dynamic spino-pelvic anomaly)
* Hip dysplasia
* Inflammatory rheumatic disease or any other progressive concomitant condition that may impact the patient's vital or functional prognosis
* Sequelae of neurological disease or stroke
* Pregnant or breastfeeding women
* Mental deficiency or any other reason that may hinder the understanding or the strict application of the protocol
* Patient likely not to return for follow-up visits
* Patient already included in another therapeutic study protocol
* Patient under court protection, guardianship or curatorship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
five-year wear thickness of the two friction pairs | Year 5
  The primary endpoint is the five-year wear thickness of the two friction pairs (CoPXE versus CoC) after total hip arthroplasty. Wear thickness is the measurement of the penetration of the femoral head into the acetabular component. This measurement will be performed on frontal pelvic radiographs centred on the pubic symphysis using the semi-automatic computer-assisted technique described by Martell

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No